CLINICAL TRIAL: NCT05196711
Title: A First-in-Human Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of MAX-40070 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety of MAX-40070 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maxinovel Pty., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAX-40070-001
Record Dates: First submitted 2021-12-07; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAX-40070 (Experimental): MAX-40070 is a liniment with two dose specification: 0.5%, 2% (Weight/Volume). In SAD phase, MAX-40070 will be applied once in each cohort, and there will be 6 cohorts. For the first 2 cohorts, 0.5% MAX-40070 will be used. For the rest 4 cohorts, 2% MAX-40070 will be used. In MAD phase, MAX-40070 2% will be applied once daily for consecutive 14 days in each cohort.
  Interventions: Drug: MAX-40070
- Placebo (Placebo Comparator): Placebo is a liniment with two dose specification: 0.5%, 2% (Weight/Volume) to match with active drug in 2:1 manner ( 6 active: 2 placebo in each cohort).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MAX-40070 — In the SAD phase, the proposed doses will be increased gradually. Each cohort will consist of 8 subjects, with 6 subjects randomly assigned to MAX-40070.
  During the MAD phase, the treatment will be administered once a day for 14 consecutive days.
  Arms: MAX-40070
Drug: Placebo — In the SAD phase, the proposed doses will be increased gradually. Each cohort will consist of 8 subjects, with 2 subjects randomly assigned to placebo
  In the MAD phase, the treatment will be administered once a day for 14 consecutive days. Each cohort will consist of 10 subjects, with 2 subjects randomly assigned to placebo
  Arms: Placebo

SUMMARY:
This is a First-in-Human phase I study to evaluate the safety, tolerability and pharmacokinetic characteristics of MAX-40070 in Healthy SubjectThe study will be comprised of 2 parts; Part A and Part B. Part A will be conducted at NZCR, and Part B will be conducted at both NZCR and another site(s) in China (if required). Part A will include approximately 48 participants, and Part B will include approximately 30 participants.

ELIGIBILITY:
Inclusion Criteria:

* Weigh at least 50kg (females) or 55kg (males) and have a BMI between 20.0 kg/m2 - 30.0 kg/m2.
* Subjects having no ulceration, damage, sunburn, redness, rash, acne, folliculitis, pigmentation, uneven skin tone, excessive freckles on the skin of the target application area and fever.

Exclusion Criteria:

* An abnormality related to the comprehensive physical examination, laboratory test, 12-lead ECG, and other diagnostic tests and which is determined by the investigator as clinically significant (CS).
* A history of CS diseases of heart, liver, lung, kidney, digestive tract, blood, or neuropsychiatric system.
* Intolerance to venipuncture for blood collection and/or having blood or needle phobia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2022-11-02 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAE) by skin irritation assessment, vital sign, ECG and clinical lab assessments | 36 Days
  skin irritation assessment will be performed during the treatment period. The dermal response score will be based on a visual irritation scale (0-7) that rates the degree of erythema, edema and other signs of cutaneous irritation. abnormal vital sign (including blood pressure, pulse rate, respiratory rate and oral temperatures), 12-lead ECG, hematology (hemoglobin, hematocrit, platelet count, RBC count, WBC count, with differential), blood chemistry (BUN, creatinine, total bilirubin, alkaline phosphatase, AST, ALT, GGT, LDH, glucose, albumin, total protein, bicarbonate, phosphate, sodium, potassium, chloride, calcium, total cholesterol, uric acid) and urinalysis (pH, specific gravity, protein, glucose, ketones, bilirubin, blood, nitrites, leukocytes, urobilinogen, microscopic urine analysis on abnormal findings) during the treatment period will be recorded and reported.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | 1 Day
  Pharmacokinetics
Time at which Cmax was first observed (Tmax) | 1 Day
  Pharmacokinetics
Area under the concentration curve from time 0 hour to 24 hour (AUC0-24) | 1 Day
  Pharmacokinetics
Area under the concentration curve for on dosing interval at steady state (AUC0-t) | 36 Days
  Pharmacokinetics

IPD SHARING:
Plan to Share IPD: Undecided